CLINICAL TRIAL: NCT04699344
Title: A Prospective, Single-centre,Single-blinded Study of PROUD for Prostate Carcinoma Diagnosis
Brief Title: A Prospective, Single-centre，Single-blinded Study of PROUD for Prostate Carcinoma Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Yueqing Tang, Principal Investigator, Qilu Hospital of Shandong University
Other Study IDs: QL-URO-001
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Prostate Carcinoma
Keywords: diagnosis
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from Urine Exfoliated Cells will be analyzed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-tissue biopsy patients: Pre-tissue biopsy patients with suspected prostate carcinoma will be the experimental group to determine the sensitivity and specificity of PROUD analysis, the result will be compared with histological results and PCA3 test.
  Interventions: Diagnostic Test: The level of CNV
- Non-cancer participants: Patients being treated for other diseases but without any tumor will provide a negative control to provide data for determining the sensitivity and specificity of PROUD analysis.
  Interventions: Diagnostic Test: The level of CNV

INTERVENTIONS:
Diagnostic Test: The level of CNV — The extracted DNA from morning urine will be analyzed by PROUD to determine the level of CNV.
  Other Names: PROUD test of the urine exfoliated cells

SUMMARY:
Prostate carcinoma (PC) is common malignancy and is considered to be the highest incidence in the old males. The traditional diagnostic methods of PC present with some shortcomings. For example, the specificity of serum PSA remains low while prostate needle biopsy is invasive and false negative in some case, even causing missed diagnosis of some high risk PC, and over diagnosis of PC is not rare. Therefore, a noninvasive diagnostic method with high accuracy is urgently needed. Our previous study has proved that PROstate cancer Urine Detector (PROUD), which is able to detect chromosomal aberrations of the urine exfoliated cells, is a reliable method in diagnosing urothelial carcinoma with sensitivity and specificity of 82.5% and 96.9%, respectively. But its potential in PC diagnosis hasn't been assessed yet and the accuracy of PROUD in detecting PC need to be validated. We here intended to investigate whether PROUD can be used in PC diagnosis and further validate the accuracy of PROUD in diagnosing PC.

DETAILED DESCRIPTION:
The traditional diagnostic methods of PC include serum PSA and prostatic biopsy (PB). To screen the PC in high risk population, PSA is commonly used. The early detection of PC is actually carried out by the association of digital rectal examination (DRE) and serum total prostate-specific antigen (tPSA) level. The usual upper limit for tPSA is 4 ng ml-1. However, between 4 and 10 ng ml-1, there exists a diagnostic grey zone with an estimated probability of only 40% of PC in men with normal findings on DRE. Prostrate cancer can only be accurately differentiated from benign prostate hyperplasia(BPH) and prostatitis by pathological proof, usually obtained by subsequent invasive PB. To refine the indications for PB, and therefore to reduce morbidity, new indicators based on tPSA were developed: age-adjusted tPSA cutoffs, tPSA velocity or tPSA density where the elevated tPSA is indexed to the gland size. The most commonly used indicator is free/total PSA ratio (f/tPSA), which may help to predict PC or BPH in its extreme values. However, the probability of PC at biopsy among men with a PSA value between 4 and 10 ng ml-1 and normal findings on DRE ranged from 56% for men with an f/tPSA ratio of <10% to 8% for men with a ratio >25%, underlying the lack of accuracy of the f/tPSA indicator. PB is the "gold standard" diagnostic procedure, which is invasive, uncomfortable and with possible adverse side effects as local bleeding and infectious complications including drug resistant bacterial strains. Furthermore, repeated tissue biopsy is needed in some cases for the missed diagnosis of PC, in the other hand, causing over diagnosis of the insignificant clinical PC cases.

The difficulty of estimating the risk of PC when there is a suspicious DRE without nodule, when tPSA ranges between 4 and 10 ng ml-1 or when f/tPSA has an average value (between 15 and 25%), taken together with the morbidity due to PB, highlights the need of new predictive markers for PC.

In urine samples, it is reported than whole-genome gene expression analysis, as noninvasive method, obtained from PC, BPH,and control groups by using the microarray system, showed the differences of gene expression profiles.To improve the specificity of prostate cancer diagnosis, prostate-cancer-specific markers, such as prostate cancer gene 3 (PCA3),are needed. The strong association between PCA3 mRNA overexpression and malignant transformation of prostate epithelium indicates its potential as a diagnostic biomarker. The PCA3 test of PC has a sensitivity ranged from 47%-69% and specificity from 72%-83%.

Copy number variations (CNVs) refers to the ongoing acquisition of genomic alterations ranging from point mutations to gross chromosomal rearrangements, is a hallmark of cancer which is found in 60-80% of human cancer, and it positively correlates with high tumor stage, poor prognosis, metastasis and therapeutic resistance. Several researches have investigated the value of detecting chromosomal instability with sWGS in either cell-free (cf)DNA or genomic DNA as a noninvasive diagnostic method for cancers and yielded quite fine results. Our previous research has also proved the PROUD model reached performance of AUC=0.928, with sensitivity, specificity and accuracy of 82.5%, 96.9% and 89.0%, respectively. This test also showed superiority in diagnosing upper tract urothelial carcinoma compared with urinary cytology test.

Here we intended to conduct a prospective, multicenter, single-blinded research to further validate the value of PROUD in diagnosing PC by analyzing the CNV level of patient DNA extracted from urine exfoliated cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected with prostate cancer and planned to undergo prostate needle biopsy.
* Patient with serum PSA test result.
* Patient willing to provide morning urine sample before biopsy, and willing to provide patient information.
* Participants without any tumor disease and willing to attend the study by providing morning urine.
* Male patients aged >= 18 years.
* Participants signed informed consent form.

Exclusion Criteria:

* Age under 18 years
* Individuals unwilling to sign the consent form or unwilling to provide morning urine for test or unwilling to provide the medical record.
* Patient already received urethral catheterization.
* Patient with late-stage uremia and need regular dialysis.
* Patient with urothelial carcinoma or suspected urothelial carcinoma.
* Suspected PC patient with endocrine therapy without histological results of the prostate.
* PC patient after any related therapy: endocrine therapy, radiotherapy, radical operation, immunotherapy, chemotherapy, transurethral prostate surgery, cryoablation or other local therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with prostate carcinoma or participants in control group from January 2021 to June 2023 in Qilu hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-25 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of urinalysis by PROUD analysis | through study completion, an average of 30 months
  number of patients "declared positive" with the PROUD test among the patients suffered from prostate cancer.
Specificity of urinalysis by PROUD analysis | through study completion, an average of 30 months
  number of patients "declared negative" with the PROUD test among the patients without cancer.
Identification of the correlation between the level of CNV and the grade (Gleason Score,GS) of the tumor sample | through study completion, an average of 30 months
  level of CNV in the urine sample compared with the grade of the tumor confirmed by histopathologic examination.
Identification of the correlation between the level of CNV and the stage (TNM) of the tumor sample. | level of CNV in the urine sample compared with the stage of the tumor confirmed by histopathologic examination.
  through study completion, an average of 30 months
Comparison of the sensitivity of the PROUD analysis versus urine PCA3 | through study completion, an average of 30 months
  number of patients "declared positive" with the PROUD analysis versus patients "declared positive" with the PCA3 test.
Comparison of the specificity of the PROUD analysis versus urine PCA3 | through study completion, an average of 30 months
  number of patients "declared negative" with the PROUD analysis versus patients " declared negative " with the PCA3 test.
Sensitivity of the PROUD analysis in different PSA subgroup(≤4,≥10，between 4-10ng ml-1) | through study completion, an average of 30 months
  number of patients "declared positive" with the PROUD test among the patients suffered from prostate cancer in different PSA subgroup(≤4,≥10，between 4-10ng ml-1).
Specificity of the PROUD analysis in different PSA subgroup(≤4,≥10，between 4-10ng ml-1). | through study completion, an average of 30 months
  number of patients "declared negative" with the PROUD test among the patients without cancer in different PSA subgroup(≤4,≥10，between 4-10ng ml-1).

CONTACTS AND LOCATIONS:
Overall Officials: Zunlin Zhou, MD, Study Chair — Qiluhospital of Shandong University
Locations (1):
- Urology Department of Qiluhospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
We will try to protect the information of the included participants

REFERENCES:
- [Result] Zeng S, Ying Y, Xing N, Wang B, Qian Z, Zhou Z, Zhang Z, Xu W, Wang H, Dai L, Gao L, Zhou T, Ji J, Xu C. Noninvasive Detection of Urothelial Carcinoma by Cost-effective Low-coverage Whole-genome Sequencing from Urine-Exfoliated Cell DNA. Clin Cancer Res. 2020 Nov 1;26(21):5646-5654. doi: 10.1158/1078-0432.CCR-20-0401. Epub 2020 Oct 9. PMID 33037018
- [Result] Thuret R, Chantrel-Groussard K, Azzouzi AR, Villette JM, Guimard S, Teillac P, Berthon P, Houlgatte A, Latil A, Cussenot O. Clinical relevance of genetic instability in prostatic cells obtained by prostatic massage in early prostate cancer. Br J Cancer. 2005 Jan 31;92(2):236-40. doi: 10.1038/sj.bjc.6602311. PMID 15655554
- [Result] Hessels D, Schalken JA. The use of PCA3 in the diagnosis of prostate cancer. Nat Rev Urol. 2009 May;6(5):255-61. doi: 10.1038/nrurol.2009.40. PMID 19424173
- [Result] Ozdemir TR, Simsir A, Onay H, Cureklibatir I, Ozkinay F, Akin H. Whole-genome gene expression analysis in urine samples of patients with prostate cancer and benign prostate hyperplasia. Urol Oncol. 2017 Oct;35(10):607.e15-607.e24. doi: 10.1016/j.urolonc.2017.05.020. Epub 2017 Jun 21. PMID 28647394